CLINICAL TRIAL: NCT05202782
Title: Phase II, Single-Arm, Open-label, Multicenter Study Evaluating the Efficacy of Adjunctive Zanubrutinib and CAR T-Cell Therapy in Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: Zanubrutinib and CAR T-cell Therapy for the Treatment of Recurrent or Refractory Aggressive B-cell Non-Hodgkin's Lymphoma or Transformed Indolent B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 20H09; NCI-2021-08866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00215064; NU 20H09 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma, Not Otherwise Specified; Large B-Cell Lymphoma With IRF4 Rearrangement; Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Recurrent Aggressive B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent Intravascular Large B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Aggressive B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory Intravascular Large B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Immunotherapy, Adoptive; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (zanubrutinib and CAR T-cell therapy) (Experimental): LEAD- IN PHASE: Patients receive zanubrutinib PO BID for 7-14 days in the absence of disease progression or unacceptable toxicity.
  CAR T-CELL THERAPY: Patients receive standard of care CAR T-cell therapy IV at 4 weeks.
  MAINTENANCE PHASE: Patients receive zanubrutinib PO BID on days 1-28. Cycles repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Zanubrutinib

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given IV
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB

SUMMARY:
This phase II trial studies the effect of zanubrutinib and CAR T-cell therapy in treating patients with aggressive B-cell non-Hodgkin's lymphoma or transformed indolent B-cell lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Zanubrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. T cells are infection fighting blood cells that can kill tumor cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize CAR, a protein on the surface of cancer cells. These CAR-specific T cells may help the body's immune system identify and kill cancer cells. Giving zanubrutinib together with CAR T-cell therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine efficacy of adjunctive zanubrutinib with chimeric antigen receptor T (CAR T)-cell therapy as defined by an improvement in 6-month complete response rates (CR) (defined per 2014 Lugano criteria) as compared to historical rates, in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) followed by maintenance zanubrutinib.

SECONDARY OBJECTIVES:

I. To determine the conversion rates of partial (PR) to complete response (CR), defined per Lugano criteria (2014), in patients with partial response to initial CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

II. To determine the overall response rate (ORR), using Lugano criteria (2014), in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

III. To determine progression free survival (PFS), in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

IV. To determine the overall survival (OS) rate in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

V. Toxicity assessment.

EXPLORATORY OBJECTIVES:

I. To determine the impact on quality of life using the health-related quality of life outcome questionnaire European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ C-30), in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

II. To measure disease-specific symptoms and/or treatment-related concerns in patients treated with CAR T-cell therapy (with a prior lead-in zanubrutinib) who are administered maintenance zanubrutinib.

III. To evaluate CAR T-cell polyfunctionality with the administration of zanubrutinib lead-in and maintenance treatment.

IV. To identify changes in immune cell subsets and cytokines with administration of zanubrutinib lead-in and maintenance.

V. To characterize potential mechanisms of loss of response by measuring changes in programmed cell death ligand-1 /2 (PD-L1/L2) and CD19 on tumor tissue.

OUTLINE:

LEAD- IN PHASE: Patients receive zanubrutinib orally (PO) twice daily (BID) for 7-14 days in the absence of disease progression or unacceptable toxicity.

CAR T-CELL THERAPY: Patients receive standard of care CAR T-cell therapy intravenously (IV) at 4 weeks.

MAINTENANCE PHASE: Patients receive zanubrutinib PO BID on days 1-28. Cycles repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histo-pathologically confirmed diagnosis of an aggressive B-cell non-Hodgkin lymphoma or transformed indolent B-cell lymphoma that is recurrent or refractory to standard therapy and with intent to treat with standard of care CAR T-cell therapy (meeting Food and Drug Administration [FDA] approved indications for the respective CAR T-cell construct being used). Standard of care /FDA approved CARTs for this population include axicabtagene ciloleucel, tisagenlecleucel or lisocabtagene maraleucel, any of which may be used for this study and provider dependent. For the purpose of this study, aggressive B-cell NHL histologies should conform to the label indications for the respective CART being utilized. Accordingly, CART eligible histologies include the following groups according to the 2016 revision of the World Health Organization (WHO) classification of lymphoid neoplasms

  * High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
  * High-grade B-cell lymphoma, not otherwise specified (NOS)
  * Diffuse large B-cell lymphoma (DLBCL), NOS
  * Diffuse large B-cell lymphoma (DLBCL), NOS; Germinal center B-cell type
  * Diffuse large B-cell lymphoma (DLBCL), NOS; Activated B-cell type
  * Large B-cell lymphoma with IRF4 rearrangement
  * T-cell/histiocyte-rich large B-cell lymphoma (subtype of DLCBL)
  * Primary cutaneous DLBCL, leg type (subtype of DLCBL)
  * Epstein-Barr virus (EBV)+ DLBCL, NOS (subtype of DLCBL)
  * DLBCL associated with chronic inflammation (subtype of DLCBL)
  * Primary mediastinal (thymic) large B-cell lymphoma
  * Intravascular large B-cell lymphoma (subtype of DLCBL)
  * Transformed indolent B-cell lymphoma; composite lymphomas with aggressive B-cell NHL as outlined above and indolent lymphomas are also allowable if felt to represent transformation
* Patients should have measurable disease per Lugano criteria (2014)
* Patients must be age >= 18 years
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have a life expectancy of greater than 12 weeks
* Females of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 500/uL neutrophil count (within 14 days of registration)
* Platelets (PLT) >= 50,000/uL (within 14 days of registration)

  * NOTE: Red blood cell (RBC) and platelet transfusion allowed >= 7 days prior to registration
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL) (within 14 days of registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (within 14 days of registration)
* Creatinine clearance >= 30 mL/min estimated by the Cockcroft-Gault equation (within 14 days of registration)
* Patients with evidence of hepatitis B virus (HBV) are eligible provided there is minimal hepatic injury and the patient has undetectable HBV on suppressive HBV therapy

  * Note: Patient must be willing to maintain adherence to HBV therapy. Patients with previously treated and eradicated hepatitis C virus (HCV) who have minimal hepatic injury are eligible
* The effects of zanubrutinib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, females of child-bearing potential (FOCBP) and men must agree to use highly effective contraception (hormonal or ; complete abstinence) from time of informed consent, for the duration of study participation, and for 180 days following completion of therapy

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
  * FOCBP must agree to practice 1 highly effective methods of contraception and 1 additional effective (barrier) method, at the same time. Otherwise females should

    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.) Females should also agree to not donate eggs (ova) during the course of this study or 180 days after receiving their last dose of study drug. Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
    * Men treated or enrolled on this protocol must also agree to use adequate contraception from time of informed consent, for the duration of study participation, and 180 days after completion of administration. Men even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following:

      * Agree to practice highly effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, OR Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
      * Agree not to donate sperm during the course of this study or 180 days after receiving their last dose of study drug.

        * Note: Female and male condoms should not be used together
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents are not eligible
* Patients who require treatment with moderate or strong CYP3A inducers =< 7 days prior to treatment with zanubrutinib lead-in are not eligible
* Patients requiring systemic treatment with corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications including anti-neoplastic therapies =< 7 days prior to treatment with zanubrutinib lead-in are not eligible

  * Please note: Steroids for treatment of lymphoma and/or management of CAR T-cell toxicities are allowed from time of apheresis until 90 days post CAR T-cell therapy. In the event that steroids are deemed necessary for CAR T-cell toxicities after 90 days, this may be done upon discussion with the principal investigator (PI)
* Patients with evidence of active disease in the central nervous system (CNS) defined as either the presence of active lesions on magnetic resonance imaging (MRI) obtained within 4 weeks prior to registration or progressive neurological decline are not eligible
* Patients are not eligible if they have uncontrolled intercurrent illness including, but not limited to

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia deemed clinically significant by the provider
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women and nursing mothers are not eligible
* Patients with human immunodeficiency virus (HIV) are not eligible
* Patients who are unable to swallow oral tablet/gel capsules are not eligible
* Patients who have gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2029-10-09 (Estimated)

PRIMARY OUTCOMES:
Change in 6-month complete response rates | At 6 months from initiation of maintenance zanubrutinib treatment
  Defined per 2014 Lugano criteria. The proportion of patients with complete response at 6 months will be estimated among evaluable of patients, and reported along with the 95% two-sided Clopper-Pearson confidence interval. A one-sample exact binomial test will be used to compare the 6-month CR rate to the historic control rate of 35%.

SECONDARY OUTCOMES:
Conversion rates of partial response (PR) to CR | At day 90, 6, 12, 18, and 24 months from initiation of zanubrutinib maintenance therapy
  Will be estimated as the proportion of patients with partial response to initial CAR T-cell therapy (following lead-in zanubrutinib) who convert to CR at any time point after initiation of zanubrutinib maintenance therapy, and will be reported as the proportion of patients who converted to CR at D90, 6, 12, 18, or 24 months, as well as at any other time point.
Overall response rate (ORR) | At day 90, 6, 12, 18, and 24 months from initiation of zanubrutinib maintenance therapy
  Assessed using Lugano criteria (2014). ORR will be defined as the percentage of patients with a CR or PR. Response will be assessed by positron emission tomography/computed tomography (CT) or CT chest/abdomen/pelvis. Will be reported using descriptive statistics.
Progression free survival | From registration until progression/recurrence of lymphoma or death from any cause, assessed at day 90, 6, 12, 18 and 24 months after initiation of zanubrutinib maintenance therapy
  Will be estimated using the method of Kaplan-Meier.
Overall survival | From registration until death from any cause, assessed at day 90, 6, 12, 18 and 24 months
  Will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | From the time of informed consent until one week post the lead- in treatment period, and then again from day 1 of maintenance treatment phase up to 30 days after treatment discontinuation
  Toxicity will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The number and percentage of toxicities will be tabulated by type, grade, severity, and attribution with each cycle of therapy. Will be summarized using descriptive statistics.

OTHER OUTCOMES:
Quality of life Questionnaire | At screening, 6 and 24 months from initiation of maintenance zanubrutinib treatment
  Assessed using health related quality of life outcome questionnaire European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30. Will be summarized using descriptive statistics.
Disease-specific symptoms and/or treatment-related concerns | At screening, 6 and 24 months from initiation of maintenance zanubrutinib treatment
  Assessed using the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy - Lymphoma Symptom lndex-18.
CAR T cell polyfunctionality | Up to 5 years
  Longitudinal analysis will be performed.
Changes in immune cell subsets and cytokines | Baseline up to 5 years
  Longitudinal analysis will be performed.
Mechanisms of loss or response | Baseline up to 5 years
  Will characterize potential mechanisms of loss or response by measuring changes in programmed cell death ligand-1 /2 (PD-L1/L2) and CD19 on tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin